CLINICAL TRIAL: NCT04237246
Title: Comparative FK506 Drug Levels of Once Daily Advagraf in First Nations and Caucasian Patients With Liver Transplants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2014:070
Record Dates: First submitted 2015-06-02; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2015-04

CONDITIONS: Liver Failure
Keywords: liver
MeSH Terms: conditions — Liver Failure | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Once daily Tacrolimus (Advegraf) (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — 24 hour "long acting" advegraf
  Other Names: Advegraf

SUMMARY:
Background:

Previous studies have documented differences in the pharmacokinetics (PK) of a once daily FK506 formulation (Advagraf) based on patient ethnicity. These findings may be of particular relevance to the First Nations population who constitute a large and increasing segment of the liver transplant population in Canada.

Aim:

The purpose of the present study is to determine whether PK differences exist for Advagraf in First Nations compared to Caucasian liver transplant patients.

Objectives:

1. Document and compare PK determinations for Advagraf in First Nations and Caucasian patients with stable liver transplants.
2. Document and compare CYP3A gene expression profiles in the two ethnic populations.

Study Design:

* single-centre, open-label
* consecutive enrollment (N=8/group)
* self-identified adult First Nations and Caucasian ethnic cohorts
* 7 day steady state conversion (mg/mg/day) from twice to once daily FK506 formulation
* timed blood samples at 0, 1.5, 2, 4, 6, and 24 hours post medication
* PK determinations:concentration at zero time (C0), time to maximum concentration (Tmax),Area Under the Curve (AUC 0-24), apparent oral clearance (CLoral) and maximum concentration (Cmax)

Methods:

* whole blood FK506 levels will be measured by UPLC tandem mass spectroscopy
* CYP3A allele analyses will be performed by Dr. Richard Kim, University of Western Ontario

Relevance:

The results of this study will serve to determine whether present guidelines for conversion of twice to once daily FK506 formulations need be modified for First Nations liver transplant patients.

DETAILED DESCRIPTION:
INTRODUCTION Immunosuppressive regimens typically include an immune modulator (e.g. azathioprine, mycophenolatemofetil or mycophenolate sodium), a steroid and a calcineurin inhibitor, either Cyclosporine or FK506. FK506 (C44H69NO12; see Figure 1) which is isolated from the fermentation broth of Streptomyces tsukubaesis2,3is a 23-membered macrolide lactone.

It is highly effective in preventing rejection in liver, kidney, heart, bone marrow, pancreas, lung and small bowel recipients and for therapy of certain autoimmune diseases4. Previous studies have documented that ethnic differences exist between the pharmacokinetic properties of FK506 given orally5-7. For example, Mancinelli et al reported that African- American (AA) transplant patients require higher FK506 dosages (mg/kg) than Asians (Chinese or Japanese) and Caucasians7. Moreover, bioavailability was significantly reduced (9.9% versus 19%) and Cmax levels were lower in AA compared to Caucasians. In a similar study, researchers in the DeKAF group6documented clinical and recipient genetic correlates of dose-normalized FK506 troughs in the first 6 months post transplant using a customized single-nucleotide polymorphism chip with 2,722 variants in a large, ethnically diverse (144 AA and 551 non-AA) adult kidney transplant population through a seven-centre consortium. In their study, AAs had consistently lower median (interquartile range) troughs than non-AAs, 6.2 (4.4-8.4) ng/mL vs 8.3 (6.4-10.4) ng/mL (P<0.0001), despite 60% higher daily doses, 8 (5-10) mg vs 5 (4-7) mg (P<0.0001). In addition, the median FK506 trough concentration at week 1 post-transplant was particularly low in AAs (2.1 [1.2-3.5] ng/mL) compared with non-AAs (5.0 [3.1-8.2] ng/mL) (P<0.0001), despite similar initial doses6.

The differences described above may result from racial differences in intestinal CYP3A or Pglycoprotein activity, since no ethnic differences were observed in the pharmacokinetics of FK506 when administrated intravenously7.CYP3A5*1 is a genotype associated with low FK506 concentrations6. However, although its effect is important, it incompletely explains the variability in FK506 concentrations and has a relatively low minor allele frequency in whites relative to AAs8,11. Nonadherence to immunosuppressive treatment is another factor that contributes to variable trough levels and potentially, adverse outcomes for various transplant populations12. Advagraf is a FK506 formulation that has been demonstrated to lower the risk of nonadherence by virtue of it being administrated once rather than twice daily5. There are an estimated 1.14 million Aboriginal peoples (largely First Nations) living in Canada with in excess of 80% residing in Ontario, British Columbia, Alberta, Manitoba and Saskatchewan. Due to a high prevalence of; viral hepatitis, non-alcoholic steatohepatitis and autoimmune chronic liver disease, First Nations peoples represent an important and increasing percentage of the country's liver transplant population13. Clinical observations in the setting of acetaminophen hepatotoxicity suggest significant differences exist in drug metabolism between the First Nations and Caucasian populations (personal communication: G.Y. Minuk). In addition, compliance with medications has been an issue in this cohort14. Thus, the present study was designed to document and compare the relative bioavailability of a once daily FK506 formulation (Advagraf) and CYP3A allele profiles in First Nations and Caucasian patients with stable liver transplants. AIM The principal aim of this study is to document and compare the oral pharmacokinetics of Tacrolimus and CYP3A allele profiles in First Nations and Caucasians with stable liver transplants. METHODS

Patients:

Study patients will be derived from the Post-Liver Transplant Clinic at the Health Sciences Centre in Winnipeg, Manitoba. At present, approximately 175 patients are being followed in the 6 December 18, 2013 clinic with 10-15% being of First Nations ethnicity. Patient ethnicity will be based on selfidentification.

Inclusion Criteria:

* First Nations or Caucasian subjects between the ages of 18 and 70 years.
* A minimum of 12 months from the transplant procedure.
* No acute rejection episode within the previous 3 months.
* No evidence of pre-transplant liver disease recurrence
* Stable Tacrolimus dosage during the previous 3 months.

Exclusion Criteria:

* Patients with absorption problems or unable to take oral medications.
* Patients who are on steroids
* Patients unable or unwilling to provide informed consent.

Pre-Study Variables:

Liver and renal function, lipid and glucose levels and arterial blood pressure determinations will be derived from the patients' last clinic visit. Liver function will have been determined by the results of liver enzyme (ALT, AST, AP and GGT) and serum bilirubin, albumin and INR values.

Renal function will be evaluated using creatinine plasma levels and by using the estimated glomerular filtration rate (GFR) derived from the Modification of Diet in Renal Disease (MDRD) equation with six variables. Patients will be defined as having renal dysfunction if the MDRD is below 60 ml/min but not excluded from the study.

Study Design:

This will be a single-centre, open-label study conducted at the Health Sciences Centre and University of Manitoba, Winnipeg, under the supervision of Drs. D. Peretz (Transplant Hepatologist) and V. Perez-Alvarez (Liver Pharmacologist). Following written informed consent, consecutively enrolled First Nations and Caucasian subjects (n=8/group) attending the Liver Transplant Outpatient Clinic at the Health Sciences Centre will receive oral FK506 capsules (mg/mg conversion, i.e. 1 mg/d of the twice daily formulation: Prograph = 1 mg/d of the once daily formulation: Advagraf) as a single daily dose for seven days until a steady state is achieved. As food has been shown to potentially interfere with the absorption of tacrolimus, patients will be NPO two hours prior to administration of the medication. On the morning of day 8, patients will be seen at the John Buhler Research Centre to begin the pharmacokinetic study. Following establishment of venous access, a baseline blood sample will be obtained. Patients will then receive Advagraf (between 8:00 and 9:00 a.m.) with 200 mL of water (T=0). Further blood sampling will be obtained at times 1.5, 2, 4 , 6 and 24 hours. The T=24 hour sample will include an additional 30 ml for subsequent CYP3A allele testing. Breakfast will be scheduled at 10:00 a.m. and a standard lunch served at 1:00 p.m.

Patients will be asked to return the following morning for the final 24 hour sample, after which they will be discharged with instructions to resume Prograph at the previous dosage (until funding for the once daily formulation is in place). Concomitant drugs will not be altered during the pharmacokinetic study. The study will be approved and monitored by the Research Ethics Board committee at the University of Manitoba and carried out according to the declaration of Helsinki and its amendments following the principles of good clinical practice. All study subjects will have provided signed informed consent, and will be free to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* First Nations or Caucasian subjects between the ages of 18 and 70 years.
* A minimum of 12 months from the transplant procedure.
* No acute rejection episode within the previous 3 months.
* No evidence of pre-transplant liver disease recurrence
* Stable Tacrolimus dosage during the previous 3 months.

Exclusion Criteria:

* Patients with absorption problems or unable to take oral medications.
* Patients who are on steroids
* Patients unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Comparative Bioavailability of a Once Daily FK506Formulation (Advagraf) in First Nations and Caucasian Patients with Stable Liver Transplants | 1 year
  pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- John Buhler Research Centre Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided